CLINICAL TRIAL: NCT05833919
Title: Second Line ERIbulin Followed by CApecitabine or the Reverse Sequence in HER2-negative Metastatic Breast Cancer (MBC) Patients: a Randomized Phase II Study - ERICA Trial
Brief Title: Second Line ERIbulin Followed by CApecitabine or the Reverse Sequence in HER2-negative Metastatic Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIM22-ERICA
Record Dates: First submitted 2023-02-01; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Capecitabine

STUDY DESIGN:
Intervention Model Description: HER 2 negative MBC patients, who have progressed to a first line chemotherapy for metastatic disease and meet all the inclusion criteria, will be considered eligible for study enrollment. Patients will be randomly allocated using a 1:1 allocation centralized method into the two study arms: ARM A or ARM B.
  Randomization will be performed with a minimization procedure that will account for the following parameters as strata:
  * center;
  * ECOG Performance Status (0-1 vs 2);
  * previous use of CDK inhibitor (yes vs no);
  * previous use of bevacizumab (yes vs no);
  * triple negative breast cancer (yes vs no).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A (Experimental): Second line Eribulin 1.23 mg/m2 i.v. on day 1, 8 every 21 days followed by third line Capecitabine 1250 mg/m2 orally twice per day on days 1 to 14 every 21 days.
  Interventions: Drug: Eribulin Mesylate; Drug: Capecitabine
- ARM B (Experimental): Second line Capecitabine 1250 mg/m2 orally twice per day on days 1 to 14 every 21 days; followed by third line Eribulin 1.23 mg/m2 i.v. on day 1, 8 every 21 days.
  Interventions: Drug: Eribulin Mesylate; Drug: Capecitabine

INTERVENTIONS:
Drug: Eribulin Mesylate — The dose of Eribulin as the ready to use solution is 1.23 mg/m2 which should be administered intravenously over 2 to 5 minutes on Days 1 and 8 of every 21-day cycle. The amount of Eribulin required (calculated above) will be withdrawn from the appropriate number of vials into a syringe. This may be injected directly as an IV bolus over 2-5 minutes or diluted in up to 100 ml 0.9% sodium chloride (NaCl) for IV infusion over 2-5 minutes.
  The dose of Eribulin may be reduced or discontinued during any cycle in accordance with the toxicity modifications described in this chapter. Toxicities will be managed by treatment interruption and dose reduction. Once the dose has been reduced, it cannot be increased at a later date
  Other Names: Eribulin
Drug: Capecitabine — Capecitabine use in breast cancer is registered as monotherapy in advanced breast cancer after failure of a taxane- and anthracycline-containing chemotherapy or for patients for whom an anthracycline is contraindicated. Capecitabine is available in tablets of 150 and 500 mg. The recommended dose as a single agent is 1,250 mg/m2 b.i.d. (twice daily) for 14 days repeated on day 22. The tablets should be swallowed with water within 30 minutes after a meal. Caution is recommended in patients with ischemic heart disease or coronary artery disease and/or in therapy with sorivudine and analogs, coumarins, and phenytoin.

SUMMARY:
GIM22-ERICA is a clinical trial investigating the efficacy of two different strategies in HER2 negative MBC treatment. The study will include MBC patients with histologically documented HER2 negative disease, who have progressed to one prior regimen for metastatic disease and are eligible for a second-line chemotherapy with either eribulin or capecitabine.

This study design should answer to different questions:

* What is the correct placement of Eribulin in the context of a long term treatment strategy?
* Is an early use of Eribulin the best approach for MBC pts treatment?
* May early use of Eribulin impact on subsequent treatment outcomes?

The correlated biomarkers analysis, evaluating angiogenic, epithelial and mesenchymal markers should confirm the results observed in preclinical studies ad support the clinical findings. Liquid biopsies and ctDNA evaluation could help to monitor the course of the disease and to identify novel biomarkers of drug resistance.

DETAILED DESCRIPTION:
Patients who are considered eligible for the study treatment, will be randomly allocated within the two study arms.

ARM A:

* Second line Eribulin 1.23 mg/m2 i.v. on day 1, 8 every 21 days
* third line Capecitabine 1250 mg/m2 orally twice per day on days 1 to 14 every 21 days

ARM B:

* Second line Capecitabine 1250 mg/m2 orally twice per day on days 1 to 14 every 21 days
* Third line Eribulin 1.23 mg/m2 i.v. on day 1, 8 every 21 days

Study treatment will be continued until disease progression, death, unacceptable toxicity, Investigator's decision or patient refusal of further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (both for clinical and blood biomarker study)
* Histological diagnosis of HER2 negative MBC
* Females ≥ 18 years
* Measurable disease (according RECIST criteria version 1.1)
* Prior Anthracyclines and Taxanes in either (neo-) adjuvant or metastatic setting, unless the patient was not suitable for one of these treatments
* 1 prior cytotoxic regimen for advanced or MBC (not including adjuvant or neo-adjuvant therapy). Patients with no prior cytotoxic regimens for advanced or metastatic disease will only be allowed if they relapsed during or within 6 months of (neo-) adjuvant cytotoxic therapy that included anathracyclines and/or taxanes (see prior criteria);
* Prior hormonotherapy and Cyclines inhibitors are allowed, so as indicated in the international guidelines for the management of hormone positive breast cancer (ER and/or PR positive);
* ECOG Performance Status ≤ 2
* Absence of angina or heart failure or infarction within 12 months from inclusion
* Adequate bone marrow and organ function as follows (haemoglobin ≥9.0 g/dl; absolute neutrophil count ≥ 1.5x103/mm3; plateled count ≥ 100x103/mm3; bilirubin levels ≤ 1.5 times Upper Limits of Normal
* biliary stenting is allowed to resolve obstruction - Serum Transaminase level ≤ 2.5 times ULN; serum creatinine ≤ 1.5 times ULN;
* Life expectancy of at least 12 weeks;
* If women of childbearing potential (WOCBP) age: effective contraceptive measures must be used during the study treatment period and up to 3 months after the last dose of study drug.

Exclusion Criteria:

* Unability to give informed consent
* Absence of measurable disease
* Concurrent active malignancies (except of in situ carcinoma of the cervix and inactive non-melanoma skin cancer)
* Current active infection;
* Serious pre-existing medical conditions or serious concomitant diseases;
* systemic disorders that would compromise the safety of the patient or her ability to complete the study, at the discretion of the investigator (for example, unstable angina pectoris, or a clinically significant history of cardiac disease or uncontrolled diabetes mellitus);
* Known immunodeficiency virus infection;
* Pregnant or breastfeeding women
* Unable to undergo medical test for geographical, social or psychological reason;
* Active or symptomatic brain metastases;
* Known complete Dihydropyrimidine dehydrogenase (DPD) deficiency (phenotype and/or genotype testing, according to applicable national guidelines, prior to the initiation of treatment with Capecitabine is recommended)
* Recent or concomitant treatment with brivudine (there must be at least a 4-week waiting period between end of treatment with brivudine and start of capecitabine therapy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Total Progression Free Survival (PFS-T) | 62 months
  Total-progression-free survival (PFS-T) is defined as the time elapsed between randomization and the first event among the following:
  * the date of progression after the second treatment on study -whichever the second treatment will be according to intention-to-treat (eventual departures from treatments planned in the protocol will be described)
  * the date of death if death occurs before second progression
  Patients who are alive and who do not fall into any of the above categories at the end of the study will be censored on the date of the last information on vital status.

SECONDARY OUTCOMES:
Overall Survival from the date of randomization | 62 months
  This is defined as the time elapsed from the first day of 2nd line therapy and death
Health-related Quality of Life (QoL) | At screening and then every 8 weeks (including at the time of disease progression/s)
  Assessment will be performed by using EORTC QoL questionnaires (QlQ C30 and specific EORTC QlQ BR23)
Disease Control Rate | 62 months
  Disease Control Rate (DCR: proportion of patients obtaining complete response or partial response or stable disease >= 6 months):
  * in second line;
  * In third line;
  * In second and/or third line.
Post Progression Survival (PPS) | 62 months
  This is defined as the time elapsed from disease progression after 3rd line of therapy and death;

OTHER OUTCOMES:
Biomarker analysis on patients' blood samples | Baseline and 62 months
  * Tumor Circulating DNA (ctDNA)
  * Angiogenetic markers (VEGF, bFGF)
  * EMT biomarkers (E- Cadherin, N-Cadherin, Vimentin, TGF-beta)
  * Leukocyte-lymphocyte subpopulations
  * Cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Mario R D'Andrea, MD, Study Chair — UOSD Oncologia, Presidio Ospedaliero San Paolo, Civitavecchia, Rome, Italy; Michelino De Laurentiis, MD, Principal Investigator — Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Naples, Italy
Locations (25):
- Italy (25):
  - Fondazione Poliambulanza, Istituto Ospedaliero, Brescia
  - A.R.N.A.S. Garibaldi - P.O. Nesima, Catania
  - A.O. Pugliese-Ciaccio, Catanzaro
  - A.O. S. Croce e Carle, Cuneo
  - Ospedale Civile degli Infermi, Faenza
  - Ospedale Fabrino Spaziani, Frosinone
  - Ospedale Policlinico San Martino, Genova
  - A.O. Ospedale Papardo, Messina
  - AORN dei Colli - Ospedale Monaldi, Napoli
  - Azienda Ospedaliero Universitaria Federico II, Napoli
  - Istituto Nazionale dei Tumori - Fondazione G. Pascale, Napoli
  - Università degli studi della Campania L. Vanvitelli, Napoli
  - P.O. Santa Maria delle Grazie - ASL Napoli 2 Nord, Pozzuoli
  - P.O. San Paolo - ASL Roma 4, Roma
  - Università Campus Biomedico, Roma
  - Policlinico Universitario Tor Vergata, Roma
  - IFO - Istituto Nazionale Tumori Regina Elena - U.O.C. Oncologia Medica 1, Roma
  - IFO - Istituto Nazionale Tumori Regina Elena - U.O.C. Oncologia Medica 2, Roma
  - Ospedale Sandro Pertini - ASL Roma 2, Roma
  - Fondazione Policlinico A. Gemelli, Roma
  - Policlinico Universitario A. Gemelli, Roma
  - Presidio Cassia Sant'Andrea - ASL Roma 1, Roma
  - ASST Lariana - Ospedale Sant'Anna, San Fermo della Battaglia
  - ASUFC P.O. "Santa Maria della Misericordia", Udine
  - ASST Sette Laghi - Ospedale Di Circolo e Fondazione Macchi, Varese

IPD SHARING:
Plan to Share IPD: No